CLINICAL TRIAL: NCT04342390
Title: Effects of High-Intensity Interval Training Exercise in Adolescents With Hepatosteatosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 260671; P20GM109096 (NIH)
Record Dates: First submitted 2020-04-08; First posted 2020-04-13 (Actual); Results first posted 2024-02-20 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2023-07

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Insulin Resistance; High Intensity Interval Training; Childhood Obesity
Keywords: NAFLD; HIIT; Insulin; Fitness; Controlled Attenuated Parameter; Steatosis; Peak oxygen uptake
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Insulin Resistance; Pediatric Obesity; Fatty Liver | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Group (Experimental): Study participants in this group will be asked to complete 4 weeks of high-intensity interval training (HIIT).
  Interventions: Other: High-Intensity Interval Training (HIIT)
- Control Group (No Intervention): Study participants in this group will not undergo HIIT exercise training during this study.

INTERVENTIONS:
Other: High-Intensity Interval Training (HIIT) — The exercise we are studying is called high-intensity interval training, or HIIT. Participants in the exercise group will participate in the exercise program. Each exercise session will last up to 1 hour. All exercise sessions will be directed and monitored by an experienced exercise trainer or exercise physiologist.
  Arms: Exercise Group

SUMMARY:
This is a research study about how short-term exercise intervention affects adolescents with a disease called non-alcoholic fatty liver disease (NAFLD).

DETAILED DESCRIPTION:
The study investigators want to learn more about the effect of a type of exercise on non-alcoholic fatty liver disease (NAFLD), and on markers of health (for example, liver, heart, and overall health) and how the body uses energy in teenagers. The exercise we are studying is called high-intensity interval training, or HIIT. Some participants in this study will receive a 4-week exercise program, and the others will not.

ELIGIBILITY:
Inclusion Criteria: Initial Enrollment

* Ages 13-18 years (inclusive) for both sexes
* Any ethnic/racial background
* English speaking competence
* Teenagers ages 13-15 weighing more than 145 pounds OR teenagers ages 16-18 weighing more than 170 pounds
* Low risk to participate in an exercise program as determined by "The Physical Activity Readiness Questionnaire for Everyone"
* Late stages of puberty (i.e., Tanner stage IV or V) based on Tanner Staging.

Inclusion Criteria: Control or Exercise Group

* Presence of Non-Alcoholic Fatty Liver Disease (NAFLD) as determined by FibroScan Controlled Attenuated Parameter (CAP) score
* Confirmed lack of diabetes as determined by Oral Glucose Tolerance Test (OGTT)
* Confirmed eligibility per medical history

Exclusion criteria:

* Pre-pubertal or early stages of puberty
* Pregnancy
* Confirmed lack of NAFLD in the past 6 months via biopsy or MRI
* Presence of an implantable medical device or metal objects in the body (a contraindication for FibroScan and/or MRI)
* High-risk to participate in an exercise program as determined by "The Physical Activity Readiness Questionnaire for Everyone"
* Unable to cooperate with study procedures and tests including genetic or physical conditions impacting mobility over the past year
* Having known chronic illnesses/disorders that may independently affect study outcome measures: type 1 diabetes mellitus, type 2 diabetes, neurologic (e.g., epilepsy), developmental (developmental delay, autism spectrum disorder), endocrine (Cushing's, growth hormone deficiency), hepatic (other than NAFLD), autoimmune, cardiac and renal disorders
* Current history of poorly-controlled asthma.
* Taking any of the following medications that can affect study outcome at the time of enrollment: insulin, metformin, or any other anti-diabetics, antipsychotics, oral steroids, and anabolic drugs (growth hormone replacement therapy, testosterone, and oxandrolone).
* Adolescents who have a history of claustrophobia.
* Adolescents who need sedation in order to complete MRI.
* Adolescents determined ineligible by the study investigator or delegated staff.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2021-04-02 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emir Tas, MD, Principal Investigator — Arkansas Children's Hospital Research Institute
Locations (2):
- United States (2):
  - Arkansas Children's Nutrition Center, Little Rock, Arkansas
  - Arkansas Children's Pediatric Clinical Research Unit, Little Rock, Arkansas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Exercise Group | Control Group
Started | 34 | 6
Completed | 31 | 6
Not Completed | 3 | 0
Not completed — Lost to Follow-up | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exercise Group | Control Group | Total
Number analyzed (Participants) | 34 | 6 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.2 (1.5) | 15.4 (1.0) | 15.2 (1.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 4 | 24
  Male | 14 | 2 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 5 | 18
  Not Hispanic or Latino | 21 | 1 | 22
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 17 | 0 | 17
  White | 17 | 6 | 23
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Intrahepatic Triglyceride (IHTG)
Description: Intrahepatic triglyceride (IHTG) percent (%) will be measured via Magnetic Resonance Imaging (MRI). IHTG percent can theoretically range between 0 and 100. By definition, an individual has Non-Alcoholic Fatty Liver Disease (NAFLD) when the IHTG percent is at or above 5 percent.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: percentage of IHTG
Arm/Group | Exercise Group | Control Group
Number analyzed (Participants) | 31 | 6
percentage of IHTG | 5.26 (3.01) | 8.97 (6.61)
Statistical Analysis 1: Comparison: Exercise Group vs Control Group; Test type: Superiority; p = 0.363, ANCOVA

2. Primary Outcome: Cardiovascular Fitness
Description: Cardiovascular fitness will be assessed via "peak oxygen uptake" (VO2 max). VO2 max is expressed as milliliters per body weight per minute in kilograms of lean body mass (mL/min/kg per LBM). There is no established normative data for VO2 max in pediatric population; however, higher values indicate better cardiovascular fitness.
Time Frame: 4 weeks
Measure: Mean (Standard Error); unit: mL/min/kg of Lean Body Mass
Arm/Group | Exercise Group | Control Group
Number analyzed (Participants) | 31 | 6
mL/min/kg of Lean Body Mass | 40.8 (7.3) | 43.2 (7.2)
Statistical Analysis 1: Comparison: Exercise Group vs Control Group; Test type: Superiority; p = 0.633, ANCOVA

3. Primary Outcome: HOMA-IR
Description: The Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) will be calculated using the fasting glucose and insulin levels. Higher HOMA-IR values indicate greater insulin resistance. HOMA-IR is calculated as "fasting insulin (microU/L) x fasting glucose (nmol/L)/22.5". HOMA-IR has an arbitrary unit. Higher numbers suggest worse outcomes.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: arbitrary unit
Arm/Group | Exercise Group | Control Group
Number analyzed (Participants) | 31 | 6
arbitrary unit | 8.69 (5.5) | 6.4 (5.5)
Statistical Analysis 1: Comparison: Exercise Group vs Control Group; Test type: Superiority; p = 0.433, ANCOVA

4. Secondary Outcome: Alanine Aminotransferase
Description: Serum alanine aminotransferase (ALT) level will be measured. ALT level is reported in international unit/liter or IU/L. Higher ALT levels suggest presence of hepatocellular damage.
Time Frame: 4 weeks
Measure: Mean (Standard Error); unit: international unit/liter
Arm/Group | Exercise Group | Control Group
Number analyzed (Participants) | 31 | 6
international unit/liter | 20.1 (17.6) | 29.7 (17.6)
Statistical Analysis 1: Comparison: Exercise Group vs Control Group; Test type: Superiority; p = 0.822, ANCOVA

5. Secondary Outcome: FibroScan - Controlled Attenuated Parameter
Description: Controlled Attenuated Parameter (CAP) score will be measured using FibroScan. CAP score is reported in decibel/meter (dB/m) and ranges between 100-400. A score of 241 dB/m or greater is consistent with non-alcoholic fatty liver disease.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: decibel/meter
Arm/Group | Exercise Group | Control Group
Number analyzed (Participants) | 31 | 6
decibel/meter | 279 (35) | 280 (35)
Statistical Analysis 1: Comparison: Exercise Group vs Control Group; Test type: Superiority; p = 0.554, ANCOVA

6. Secondary Outcome: FibroScan - Transient Elastogram
Description: Transient Elastogram (TE) score will be measured using FibroScan. TE score is reported in kilopascals (kPa) and ranges between 0-75. A score of 8.5 kPa or greater is consistent with fibrotic liver disease.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: kPa
Arm/Group | Exercise Group | Control Group
Number analyzed (Participants) | 31 | 6
kPa | 5 (1) | 5 (3)
Statistical Analysis 1: Comparison: Exercise Group vs Control Group; Test type: Superiority; p = 0.186, ANCOVA

7. Secondary Outcome: Body Composition - Total Body Fat
Description: Body composition will be measured using Dual X-Ray Absorptiometry (DXA) scan. Normative data for total body fat is not established; however, larger total body fat percentage (percentage of total body weight) is linked to higher intrahepatic triglyceride content and insulin resistant state.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: percentage of total body weight
Arm/Group | Exercise Group | Control Group
Number analyzed (Participants) | 31 | 6
percentage of total body weight | 45.35 (6.18) | 44.05 (6.18)
Statistical Analysis 1: Comparison: Exercise Group vs Control Group; Test type: Superiority; p = 0.921, ANCOVA

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Exercise Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/6
Other Adverse Events (participants affected / at risk) | 1/34 | 0/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exercise Group (N=34) | Control Group (N=6)
muscle sprain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-16): https://cdn.clinicaltrials.gov/large-docs/90/NCT04342390/Prot_SAP_000.pdf